CLINICAL TRIAL: NCT02303743
Title: Improving the Quality of Colonoscopy Bowel Preparation Using a Smart Phone Application
Brief Title: Improving Bowel Cleansing With a Smart Phone Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vicente Lorenzo-Zúñiga García (Other)
Responsible Party: Sponsor-Investigator, Vicente Lorenzo-Zúñiga García, M.D.; Ph.D., Germans Trias i Pujol Hospital
Organization: Germans Trias i Pujol Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEI071114
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2015-01

CONDITIONS: Cathartics; Mobile Applications
Keywords: Bowel preparation; colonoscopy; Smartphone application

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smart Phone Application (SPA) Group (Active Comparator): Patients assigned to SPA group were instructed on how to free-download the application onto their smartphone. Each patient enters the date and time of his colonoscopy and timed alerts appeared on the phone to alert the patient of the next step in bowel preparation. In addition to the alerts, the app assists in bowel preparation by explaining the procedure, providing tips, examples of low fiber diet, and displaying pictures of preparation quality and educational video to explain how to prepare the purgative solution.Finally, the patient can obtain a checklist to confirm all steps.
  Interventions: Device: Smart Phone Application
- Control Group (Active Comparator): Written instructions with visual aids explaining the procedure and when to begin self-administration of the bowel solution
  Interventions: Device: Written instructions with visual aids

INTERVENTIONS:
Device: Smart Phone Application — Bowel preparation was evaluated using the Harefield Cleansing Scale (HCS). The scale was the primary outcome measure
  Arms: Smart Phone Application (SPA) Group
Device: Written instructions with visual aids — written instructions with visual aids explaining the procedure and when to begin self-administration of the bowel solution (control group).
  Arms: Control Group

SUMMARY:
Getting ready for a colonoscopy is difficult and involves a lot of steps. The information given to patients is very important to adherence to treatment. The investigators have created a novel smart phone application (SPA) aimed to increased bowel preparation quality and patient satisfaction, using different educational tools.

DETAILED DESCRIPTION:
Background: Getting ready for a colonoscopy is difficult and involves a lot of steps. The information given to patients is very important to adherence to treatment. The investigators have created a novel smart phone application (SPA) aimed to increased bowel preparation quality and patient satisfaction, using different educational tools.

Methods: The investigators have performed a prospective, endoscopist-blinded, randomized, controlled trial. The investigators have enrolled 260 outpatients owners of a smartphone. Patients were randomly allocated to two different protocols: instructions provided by SPA (SPA group; n=108) or written instructions with visual aids (control group; n=152). All procedures were performed in afternoon time and patients received the same purgative regimen (2-L PEG solution plus ascorbic acid), in a full-dose same-day regimen. The day before colonoscopy (Baseline), patients initiated low fiber diet. The study was designed to detect an improvement in quality of bowel preparation using the Harefield Cleansing Scale (HCS) scale. The effect of protocol on patient satisfaction was assessed with a specific questionnaire at time of the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Elective colonoscopy
* Owners of a smartphone

Exclusion Criteria:

* No owners of a smartphone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Lorenzo-Zúñiga Garcíaa, M.D.; Ph.D., Principal Investigator — Germans Trias i Pujol Hospital

REFERENCES:
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Spiegel BM, Talley J, Shekelle P, Agarwal N, Snyder B, Bolus R, Kurzbard N, Chan M, Ho A, Kaneshiro M, Cordasco K, Cohen H. Development and validation of a novel patient educational booklet to enhance colonoscopy preparation. Am J Gastroenterol. 2011 May;106(5):875-83. doi: 10.1038/ajg.2011.75. Epub 2011 Apr 12. PMID 21483463
- [Background] Tae JW, Lee JC, Hong SJ, Han JP, Lee YH, Chung JH, Yoon HG, Ko BM, Cho JY, Lee JS, Lee MS. Impact of patient education with cartoon visual aids on the quality of bowel preparation for colonoscopy. Gastrointest Endosc. 2012 Oct;76(4):804-11. doi: 10.1016/j.gie.2012.05.026. Epub 2012 Jul 27. PMID 22840295
- [Background] Prakash SR, Verma S, McGowan J, Smith BE, Shroff A, Gibson GH, Cheng M, Lowe Ii D, Gopal K, Mohanty SR. Improving the quality of colonoscopy bowel preparation using an educational video. Can J Gastroenterol. 2013 Dec;27(12):696-700. doi: 10.1155/2013/292636. PMID 24340313
- See also: Moviprep: ASCORBIC ACID; POLYETHYLENE GLYCOL 3350; POTASSIUM CHLORIDE; SODIUM ASCORBATE; SODIUM CHLORIDE; SODIUM SULFATE — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&DrugName=MOVIPREP&CFID=1139220&CFTOKEN=5edcdf6f70d014fa-11A89A4A-EB21-994E-AFC340D177A37A92

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smart Phone Application (SPA) Group | Control Group
Started | 108 | 152
Completed | 108 | 152
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Men and women aged 18 and older with scheduled elective colonoscopy. All enrolled outpatients were able to follow instructions and owners of a smartphone
Groups:
- Total: Total of all reporting groups
Arm/Group | Smart Phone Application (SPA) Group | Control Group | Total
Number analyzed (Participants) | 108 | 152 | 260
Age, Continuous [Mean (Full Range); unit: years] | 48 [30 to 66] | 52 [21 to 85] | 50 [21 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 100 | 160
  Male | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Bowel Preparation Was Evaluated Using the Harefield Cleansing Scale (HCS). The Scale Was the Primary Outcome Measure
Description: The quality of bowel cleansing is evaluated after colonoscopy (Day 1). Baseline the patients initiated low fiber diet in the 24 hours prior to colonoscopy. The HCS uses a 5-point qualitative scale in 5 separate colon segments. HCS is the sum of 5 segments, ranging from 0 (worst possible outcome) to 20 (best possible outcome). Global score assesses the quality of bowel cleansing: Successful (A or B) / unsuccessful (C or D). A: All segments scored 3 or 4; B: One or more segments scored 2; C: One or more segments scored 1; and D: One or more segments scored 0.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smart Phone Application (SPA) Group | Control Group
Number analyzed (Participants) | 108 | 152
units on a scale | 17.05 (3.2) | 16.52 (3.1)

2. Secondary Outcome: Patient Satisfaction Were Assessed With a Specific Questionnaire
Description: Patient satisfaction were assessed with a specific questionnaire before colonoscopy. Patients were asked if they used the application and their satisfaction with the app. Again, the endoscopist was blinded to the answers. The items read as follows: (1) "Do you have experience with a previous colonoscopy?"; (2) "Have you used the phone application?"; (3) "How easy was the preparation for colonoscopy?"; (4) "Which is your level of satisfaction with the bowel preparation?"; (5) "Would you like to repeat the same preparation in the future?"; (6) "Did you have any difficulty with the preparation?". Patient responses to the questionnaire were categorical (yes or no; questions 1, 2, 5, and 6) or numerical scale answers (0 to 10), from very difficult or very bad (0 or close to 0) to very easy or very good (10 or close to 10) (items 3 and 4).
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smart Phone Application (SPA) Group | Control Group
Number analyzed (Participants) | 108 | 152
units on a scale
  Level of satisfaction (Range 0 to 10) | 8.7 (1.6) | 6.9 (2.7)
  Ease of preparation for colonoscopy (Range 0 to 10 | 8.4 (1.7) | 7.8 (2.0)

ADVERSE EVENTS:
Time Frame: 6 months (from January to June 2014).
Description: Other (Not Including Serious) Adverse Events were not collected for any participants
Arm/Group | Smart Phone Application (SPA) Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/152
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes